CLINICAL TRIAL: NCT05712772
Title: Neuro-affective Response to Light in Depressed Adolescents and Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Adriane Soehner, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY22040093; R21MH127294 (NIH)
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Depression in Adolescence; Depression in Adults
MeSH Terms: interventions — Blue Light; Red Light

STUDY DESIGN:
Intervention Model Description: All participants will receive blue and red light exposures; order of red vs. blue light will be counterbalanced across participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blue then Red Light (Experimental): Blue light (480 nm) then Red light (640 nm)
  Interventions: Other: Blue Light; Other: Red Light
- Red Light then Blue Light (Experimental): Red light (640 nm) then Blue light (480 nm)
  Interventions: Other: Blue Light; Other: Red Light

INTERVENTIONS:
Other: Blue Light — Blue light exposure
Other: Red Light — Red light exposure

SUMMARY:
The goal of this neuroimaging pilot study is to understand developmental differences in the impact of therapeutic wavelength light (blue light) versus a non-therapeutic wavelength (red light) on emotional brain function in depression. The main questions this study aims to answer are:

* Does acute exposure to blue light (vs red light) stabilize emotional brain function in depressed individuals?
* Are stabilizing effects of blue light (vs red light) stronger for blue light in adolescents than young adults?

Participants will complete:

* A magnetic resonance imaging brain scan, in which we will examine the effect of blue versus red light on emotional brain function at rest and in response to rewards and losses.
* A pupillometry test of sensitivity to blue vs red light
* Clinical interviews and surveys
* Screening measures for drug and alcohol use, MRI safety, and current pregnancy [if relevant]
* Home sleep tracking with sleep diary and actigraphy for one week

ELIGIBILITY:
Inclusion Criteria:

* Elevated Depressive Symptoms [PHQ9≥5 And (Item 1≥1 or Item 2≥1)]
* (If <18yr) Parent or guardian can attend the baseline clinical interview

Exclusion Criteria:

* Unable to read and write in English
* Intellectual disability.
* Left or mixed handedness
* Changes to psychotropic medication type or dosage in the past 2 months
* Lifetime bipolar disorder or schizophrenia, or substance/alcohol disorder in the past 3 months.
* Factors influencing light and color sensitivity (i.e., color-blindness, serious ophthalmological conditions, photo-sensitizing medication).
* Factors influencing the ability to maintain a stable sleep schedule (i.e., shift work, severe sleep disorders, extremely late or early sleep schedule).
* Severe medical illness, neurological disorders, or history of head trauma.
* Current pregnancy or nursing
* MRI contraindication (e.g., metals in the body, recent tattoo, claustrophobia)
* Positive alcohol or substance use screen at MRI visit

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Amygdala cerebral blood flow during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  Cerebral blood flow will be assessed using pseudo-continuous arterial spin labeling collected during blue and red light exposures. Regional cerebral blood flow in the amygdala region of interest will be examined.
Ventral Striatum cerebral blood flow during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  Cerebral blood flow will be assessed using pseudo-continuous arterial spin labeling collected during blue and red light exposures. Regional cerebral blood flow in the ventral striatum region of interest will be examined.
Amygdala activity (loss>neutral) during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  This outcome will be measured during the an auditory probabilistic reward task, which is a computerized fMRI behavioral task. Activation is defined by blood oxygen dependent signal within an amygdala region of interest on loss versus neutral (no win/no loss) trials.
Ventral Striatum activity (punish>neutral) during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  This outcome will be measured during the an auditory probabilistic reward task, which is a computerized fMRI behavioral task. Activation is defined by blood oxygen dependent signal within a ventral striatum region of interest on win versus neutral (no win/no loss) trials.

SECONDARY OUTCOMES:
Medial prefrontal cortex cerebral blood flow during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  Cerebral blood flow will be assessed using pseudo-continuous arterial spin labeling collected during blue and red light exposures. Regional cerebral blood flow in the medial prefrontal region of interest will be examined.
Insula cerebral blood flow during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  Cerebral blood flow will be assessed using pseudo-continuous arterial spin labeling collected during blue and red light exposures. Regional cerebral blood flow in the insula regions of interest will be examined.
Ventromedial prefrontal cortex cerebral blood flow during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  Cerebral blood flow will be assessed using pseudo-continuous arterial spin labeling collected during blue and red light exposures. Regional cerebral blood flow in the ventromedial prefrontal cortex regions of interest will be examined.
Amygdala-whole brain functional connectivity (loss>neutral) during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  This outcome will be measured during the an auditory probabilistic reward task, which is a computerized fMRI behavioral task. Functional connectivity is defined as a psychophysiological interaction between the seed region (amygdala) and the whole brain on loss versus neutral (no win/no loss) trials
Ventromedial prefrontal cortex activity (loss>neutral) during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  This outcome will be measured during the an auditory probabilistic reward task, which is a computerized fMRI behavioral task. Activation is defined by blood oxygen dependent signal within the ventromedial prefrontal cortex region of interest on loss versus neutral (no win/no loss) trials.
Insula activity (loss>neutral) during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  This outcome will be measured during the an auditory probabilistic reward task, which is a computerized fMRI behavioral task. Activation is defined by blood oxygen dependent signal within the insula region of interest on loss versus neutral (no win/no loss) trials.
Medial prefrontal cortex activity (win>neutral) during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  This outcome will be measured during the an auditory probabilistic reward task, which is a computerized fMRI behavioral task. Activation is defined by blood oxygen dependent signal within the medial prefrontal region of interest on win versus neutral (no win/no loss) trials.
Ventral striatum-whole brain functional connectivity (win>neutral) during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  This outcome will be measured during the an auditory probabilistic reward task, which is a computerized fMRI behavioral task. Functional connectivity is defined as a psychophysiological interaction between the seed region (ventral striatum) and the whole brain.
Ventromedial prefrontal cortex activity, insula, and medial prefrontal activity, and amygdala- and ventral striatum whole brain functional connectivity (response bias; B') during Blue vs Red light exposure | Collected during the blue and red light exposures during the MRI scan at the lab visit
  This outcome will be measured during the an auditory probabilistic reward task, which is a computerized fMRI behavioral task. Activation is defined by blood oxygen dependent signal within the above regions of interest using a response bias metric (B'). Functional connectivity is defined as a psychophysiological interaction between the seed regions (amygdala, ventral striatums) and the whole brain.

CONTACTS AND LOCATIONS:
Overall Officials: Adriane M Soehner, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will complete and submit a National Data Archive (NDA) Data Sharing Agreement within 6 months of the Notice of Award Issue date. Study staff will upload data dictionary to the NDA website, and will review the NDA data definition for the measures collected and define the project's data definition harmonized to that standard. For measures not yet defined, project staff will work with the NDA staff to define the measure following NDA best practices. Informed consent will be collected from study participants that allows for broad sharing of participants' de-identified data. Study staff will use participants' personally identifiable information to generate NDA Global Unique Identifier (GUID) numbers for study participants.
  All data will be identified by GUID numbers only prior to submission to the NDA database. Data transfer procedures will be in accordance with all Institutional Review Board guidelines and federal regulations including HIPAA.
Time Frame: Raw data and data from descriptive/raw measures will be submitted on a semi-annual basis by July 15 and January 15 or the next business day. We also agree to submit to NDA the analyzed data yielded in our project (i.e., 12 months after accomplishment of each primary aim or objective, or immediately upon publication of the project's primary results, whichever occurs first). The PIs reserve the right to publish on the stated aims in a timely manner during the period of the award. Data will be available for addressing other research questions (i.e. which are not described in funded/pending grants) as soon as the data have been checked for accuracy (a period which will be no later than one year after the completion of each assessment). After the award has ended, the study investigators will continue to test the stated aims, but will also continue to solicit collaborations with outside researchers and to consider data requests in a timely manner.
Access Criteria: Outside investigators must submit a 1) proposal of the study aims, hypotheses, variables/constructs, analytic approach, and estimated duration of the proposed research; 2) resume, qualifications, source of financial support, and conflict of interest statement; 3)sign a data-sharing agreement and confidentiality statement that stipulates using the data for the stated research purposes only, securing the data using appropriate computer technology, not manipulating the data in order to identify participants, acknowledging the grant that supported data collection and management in publications/presentations, and destroying or returning the data after analyses are complete; 4) obtain approval from their Institutional Review Board, and along with other staff members who have access to the data, submit certificates of human subjects protection training.
URL: https://nda.nih.gov/